CLINICAL TRIAL: NCT03776084
Title: Evaluation of Compliance With CPAP Therapy in Patients Diagnosed With Obstructive Sleep Apnea Syndrome at the Hospital de Sabadell
Brief Title: Compliance With Continuous Positive Airway Pressure Therapy in Patients With Obstructive Sleep Apnea Syndrome
Acronym: CPAPSH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Montserrat Montaña, Principal Investigator, Clinical Research, Corporacion Parc Tauli
Other Study IDs: 2018569
Record Dates: First submitted 2018-12-13; First posted 2018-12-14 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Sleep Apnea, Obstructive
Keywords: treatment adherence and compliance; attitudes; Continuous Positive Airway Pressure; cross-cultural validation
MeSH Terms: conditions — Sleep Apnea, Obstructive; Treatment Adherence and Compliance; Behavior | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients SAHS with CPAP: Continuous Positive Airway Pressure treatment
  Interventions: Device: Continuous Positive Airway Pressure

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — CPAP indication

SUMMARY:
The aim of the study is to know the adherence to treatment and compliance of patients diagnosed with SAHS and with indication of CPAP from the sleep unit of the Hospital de Sabadell.

DETAILED DESCRIPTION:
The investigatror's objective will be to know the adherence to treatment and compliance of patients diagnosed with SAHS and with indication of CPAP of the sleep unit of the Hospital de Sabadell. Is a cohort study. The dependent variables are adherence to treatment (% patients who continue using CPAP one year after initiation of treatment) and objective compliance with treatment (defined as use of ≥4h / night). For a confidence level of 95%, a sample of 405 patients was recruited, recruited consecutively at a rate of 33 patients per month among those diagnosed with SAHS and those indicated with CPAP treatment. This number foresees a possible abandonment rate of 5%. For the statistical analysis of the data related to compliance with the therapy and compliance with the follow-up process, descriptive analysis of the data with means, median and 95% CI, or percentages with 95% CI. For the statistical analysis of the factors influencing compliance: multivariate logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age treated with CPAP based on the diagnosis of OSAS (clinical picture and AHI> 10).

Exclusion Criteria:

* Diagnosis of a psychiatric illness or dementia.
* Communication problems or inability to read and speak Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with OSAS and who underwent treatment with Continuous Positive Airway Pressure at the Hospital de Sabadell.
Sampling Method: Non-Probability Sample
Enrollment: 405 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Adherence rate to CPAP treatment | 1 year after starting treatment
  % of patients who still use CPAP
Ratio of patients with compliance with the treatment | 1 year after starting treatment
  % of patients use CPAP ≥4h / night

CONTACTS AND LOCATIONS:
Overall Officials: Montserrat Montaña, PHD, Principal Investigator — Corporacion Parc Tauli
Locations (1):
- CorporacionPT, Sabadell, Barcelona, Spain